CLINICAL TRIAL: NCT04772027
Title: Characterization and Identification of Motor Parameters Using Instrumental Assessment in Patients With Limb Girdle Muscular Dystrophy
Brief Title: Motor Parameters in Patients With Limb Girdle Muscular Dystrophy
Acronym: EIDY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200141; 2020-A02090-39 (Registry Identifier: IDRCB)
Record Dates: First submitted 2021-01-07; First posted 2021-02-25 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Limb Girdle Muscular Dystrophies
Keywords: Limb Girdle Muscular Dystrophies (LGMD); motricity; instrumental assessment
MeSH Terms: conditions — Muscular Dystrophies, Limb-Girdle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Muscular dystrophies group: 40 patients with limb girdle muscular dystrophie
- Comparator group: 40 healthy volunteers without neuromuscular or squeletic disorder

SUMMARY:
The primary objective of the study is to perform 2-year follow up with motor parameters evolution using instrumental assessments in patients with limb girdle muscular dystrophie, and to identify which motor parameters are sensitive to change.

The secondary objectives of the study are:

* to describe the changes of the parameters obtained from instrumental evaluations in comparison with the changes obtained from clinical assessments.
* to characterize the muscular impairments, the biomechanical gait disorders, the standing postural control disorders, the biomechanical upper limb disorders in spatial exploration, the limitation of upper limb capacities, the fatigue, the endurance, the patients' participation to their activities and their quality of life, in comparison with a healthy paired population.
* to highlight the relationships between muscular assessment parameters, biomechanical gait parameters, standing posture control and upper limb spatial exploration.
* to highlight the relationships between data from instrumental assessments and data from clinical assessments.
* to highlight the relationships between instrumental assessments data and clinical assessments data on one side, and features of patients (age, sex, duration since diagnosis, type of LGMD, rehabilitation in follow-up, sportive practices...) on the other side.

DETAILED DESCRIPTION:
This is a monocentric study in which 2 sub-groups of people will be enrolled: LGMD patients and healthy volunteers. Each enrolled LGMD patient will have 5 visits during 2 years, one baseline visit and four half-yearly visits. Each enrolled healthy volunteer will have one planned visit only. The duration of enrollments will last 20 months.

ELIGIBILITY:
Inclusion Criteria:

* For limb girdle muscular dystrophie group:

  * Patients diagnosed limb girdle muscular dystrophie;
  * Aged between 18 and 70 years;
  * Covered by the French social security scheme;
  * Patient able to maintain upright position alone;
  * Able to walk at least 10 meters and 6 minutes consecutively without help.
* For Volunteer group:

  * Adult (18 to 70 years) without neuromuscular or squeletic disorder.

Exclusion Criteria:

§ For all:

* Without associated neuromuscular disorders such as respiratory or muscular-squeletic diseases, apart from the consequences of dystrophy;
* Contraindication to the tests;
* Noncontrol cardiac rhythm disorders;
* Lying down position intolerance due to severe respiratory troubles;
* Pregnant or breastfeeding woman.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population with limb girdle muscular dystrophie for 2-year longitudinal follow-up in Raymond Poincaré hospital. The 4 most common types of diseases: calpainopathy, sarcoglycanopathy, dysferlinopathy and alpha-dystroglycanopathy.
  Control group: healthy population without neuromuscular or squeletic disorder.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline on maximal strength | Assessed at 6 months, 12 months, 18 months and 24 months
  Maximal strength and muscular activation of knee extensors will be evaluated by isometric test with an isokinetic dynamometer (Biodex Medical Systems Inc., Shirley, New York, USA).
Change from baseline on peak hip flexion | Assessed at 6 months, 12 months, 18 months and 24 months
  Hip flexion peak during gait will be evaluated with tridimensional gait analysis with an optoelectronic system ((Optitrack system, Natural Point Inc. Corvallis, OR, USA)
Change from baseline on speed of center of pression during standing postural control | Assessed at 6 months, 12 months, 18 months and 24 months
  Speed of center of pression will be measured by force platforms (AMTI, Advanced Mechanical Technology).
Change from baseline on elbow peak extension during upper limb spatial exploration | Assessed at 6 months, 12 months, 18 months and 24 months
  Elbow peak extension will be measured biomechanically with an optoelectronic system during upper limb spatial exploration (Optitrack system, Natural Point Inc. Corvallis, OR, USA)

SECONDARY OUTCOMES:
Change from baseline on muscular parameters | Assessed at 6 months, 12 months, 18 months and 24 months
  Maximal strength during isometric tests of hip, knee flexors, ankle and maximal grip strength. (Biodex Medical Systems Inc., Shirley, New York, USA) Muscular fatigue
Joint kinematic parameters: change from baseline on gait speed | Assessed at 6 months, 12 months, 18 months and 24 months
  Spatio-temporal from biomechanical gait analysis: an optoelectronic system (Optitrack system, Natural Point Inc. Corvallis, OR, USA) will be used.
  Spatio-temporal = speed (m/s)
Joint kinematic parameters: change from baseline on step length | Assessed at 6 months, 12 months, 18 months and 24 months
  Spatio-temporal from biomechanical gait analysis: an optoelectronic system (Optitrack system, Natural Point Inc. Corvallis, OR, USA) will be used.
Joint kinematic parameters: change from baseline on cadence | Assessed at 6 months, 12 months, 18 months and 24 months
  Spatio-temporal from biomechanical gait analysis: an optoelectronic system (Optitrack system, Natural Point Inc. Corvallis, OR, USA) will be used.
Joint kinematic parameters: change from baseline on step width | Assessed at 6 months, 12 months, 18 months and 24 months
  Spatio-temporal from biomechanical gait analysis: an optoelectronic system (Optitrack system, Natural Point Inc. Corvallis, OR, USA) will be used.
Joint kinematic parameters: change from baseline on % single support phase of gait cycle | Assessed at 6 months, 12 months, 18 months and 24 months
  Spatio-temporal from biomechanical gait analysis: an optoelectronic system (Optitrack system, Natural Point Inc. Corvallis, OR, USA) will be used.
Joint kinematic parameters: change from baseline on % swing phase of gait cycle | Assessed at 6 months, 12 months, 18 months and 24 months
  Spatio-temporal from biomechanical gait analysis: an optoelectronic system (Optitrack system, Natural Point Inc. Corvallis, OR, USA) will be used.
Joint kinematic parameters: change from baseline on % support phase of gait cycle | Assessed at 6 months, 12 months, 18 months and 24 months
  Spatio-temporal from biomechanical gait analysis: an optoelectronic system (Optitrack system, Natural Point Inc. Corvallis, OR, USA) will be used.
Change from baseline on kinetic gait parameters | Assessed at 6 months, 12 months, 18 months and 24 months
  Kinetic parameters will be obtained from biomechanical gait analysis with AMTI force plateforms (Advanced Mechanical Technology, Waterton, MA, USA).
  This includes peak of ground reaction force in antero-posterior and vertical axis.
Change from baseline on standing postural control parameters: COP displacements | Assessed at 6 months, 12 months, 18 months and 24 months
  Parameters of stabilization and postural orientation during postural control assessment on force platforms (AMTI, Advanced Mechanical Technology), Waterton, MA, USA). Parameters of stabilization include:
  Mean and maximal speed of center of pression (COP) displacements.
Change from baseline on standing postural control parameters: elliptic surface | Assessed at 6 months, 12 months, 18 months and 24 months
  Parameters of stabilization and postural orientation during postural control assessment on force platforms (AMTI, Advanced Mechanical Technology), Waterton, MA, USA). Parameters of stabilization include:
  Elliptic surface covering 90% of COP positions.
Change from baseline on standing postural control parameters: Amplitude of COP | Assessed at 6 months, 12 months, 18 months and 24 months
  Parameters of stabilization and postural orientation during postural control assessment on force platforms (AMTI, Advanced Mechanical Technology), Waterton, MA, USA). Parameters of stabilization include:
  Amplitude of COP shift in anteroposterior and mediolateral axis.
Change from baseline on standing postural control parameters: Romberg quotient | Assessed at 6 months, 12 months, 18 months and 24 months
  Parameters of stabilization and postural orientation during postural control assessment on force platforms (AMTI, Advanced Mechanical Technology), Waterton, MA, USA). Parameters of stabilization include:
  Romberg quotient.
Change from baseline on standing postural orientation parameters | Assessed at 6 months, 12 months, 18 months and 24 months
  Parameters of stabilization and postural orientation during postural control assessment on force platforms (AMTI, Advanced Mechanical Technology), Waterton, MA, USA).
  The orientation parameters include: mean position of COP in anteroposterior and mediolateral axis.
Change from baseline on standing postural orientation parameters: limb loading ratio | Assessed at 6 months, 12 months, 18 months and 24 months
  Parameters of stabilization and postural orientation during postural control assessment on force platforms (AMTI, Advanced Mechanical Technology), Waterton, MA, USA).
  The orientation parameters include: limb loading ratio.
Change from baseline on drinking task with left and right upper limb: velocity and movement time | Assessed at 6 months, 12 months, 18 months and 24 months
  The spatio-temporal parameters will be obtained from biomechanical analysis with an optoelectronic system (Optitrack system, Natural Point Inc. Corvallis, OR, USA) including:
  Velocity and movement time (Total movement time / Peak velocity/ Mean velocity)
Change from baseline on drinking task with left and right upper limb: movement strategy | Assessed at 6 months, 12 months, 18 months and 24 months
  The spatio-temporal parameters will be obtained from biomechanical analysis with an optoelectronic system (Optitrack system, Natural Point Inc. Corvallis, OR, USA) including:
  Movement strategy (Time to peak velocity / time to first peak)
Change from baseline on drinking task with left and right upper limb: smoothness and coordination movement | Assessed at 6 months, 12 months, 18 months and 24 months
  The spatio-temporal parameters will be obtained from biomechanical analysis with an optoelectronic system (Optitrack system, Natural Point Inc. Corvallis, OR, USA) including:
  Smoothness and coordination movement (number of movements units / interjoint coordination)
Change from baseline on drinking task with left and right upper limb: trunk displacement | Assessed at 6 months, 12 months, 18 months and 24 months
  The spatio-temporal parameters will be obtained from biomechanical analysis with an optoelectronic system (Optitrack system, Natural Point Inc. Corvallis, OR, USA) including:
  Trunk displacement
Change from baseline on drinking task with left and right upper limb: angular joint | Assessed at 6 months, 12 months, 18 months and 24 months
  The spatio-temporal parameters will be obtained from biomechanical analysis with an optoelectronic system (Optitrack system, Natural Point Inc. Corvallis, OR, USA) including:
  Angular joint
Change from baseline on 6 minutes walking test distance | Assessed at 6 months, 12 months, 18 months and 24 months
  6 minutes walking test
Change from baseline on the Berg Balance Scale score | Assessed at 6 months, 12 months, 18 months and 24 months
  The Berg Balance Scale
Change from baseline on Brooke Upper Extremity Scale score | Assessed at 6 months, 12 months, 18 months and 24 months
  Brooke Upper Extremity Scale score for upper extremity capacities.
Change from baseline on locomotor | Assessed at 6 months, 12 months, 18 months and 24 months
  Questionnaires Abiloco
Change from baseline on upper limb capacities | Assessed at 6 months, 12 months, 18 months and 24 months
  Questionnaires Abilhand
Change from baseline on patient occupations | Assessed at 6 months, 12 months, 18 months and 24 months
  Patient occupations assessed by COPM (Canadian Occupational Performance Measure). The measurement will be from 1 (not at all performant) to 10 (very performant) as score.
Change from baseline on MRC (Medical Research Council) score on flexors and extensors of lower and upper limb | Assessed at 6 months, 12 months, 18 months and 24 months
  Testing MRC (Medical Research Council), a scale for muscle power. The muscle scale grades muscle power on a scale of 0 to 5 in relation to the maximum expected for that muscle.
Change from baseline on Fatigue Severity Scale (FSS) score | Assessed at 6 months, 12 months, 18 months and 24 months
  Questionnaire Fatigue Severity Scale (FSS) for fatigue assessment
Change from baseline on number of fall risks | Assessed at 6 months, 12 months, 18 months and 24 months
Change from baseline on number of physiotherapy sessions per week | at baseline, 6 months, 12 months, 18 months and 24 months
Change from baseline on number of sports practice per week | at baseline, 6 months, 12 months, 18 months and 24 months
Change from baseline on Individualized Neuromuscular Quality of Life Questionnaire (INQoL) | Assessed at 6 months, 12 months, 18 months and 24 months
  Quality of life questionnaire: INQoL

CONTACTS AND LOCATIONS:
Overall Officials: Céline BONNYAUD, PhD, Principal Investigator — Laboratoire d'analyse du mouvement, Service d'explorations fonctionnelles, Hôpital Raymond Poincaré, APHP; Samuel POUPLIN, Study Director — Plateforme Nouvelles Technologies, Hôpital Raymond Poincaré, APHP
Locations (1):
- Laboratoire d'analyse du mouvement, Service d'exploration fonctionnelles, Hôpital Raymond Poincaré, APHP, Garche, France

IPD SHARING:
Plan to Share IPD: No